CLINICAL TRIAL: NCT06407297
Title: Investigation of Dose Escalation and Cohort Expansion Study on the Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells(UCMSCs) Combined With Standard Therapy for Newly Diagnosed Type 1 Diabetes
Brief Title: UCMSCs Combined With Standard Therapy for the Treatment of Newly Diagnosed Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZYZ-T1DM-2023-IIT
Record Dates: First submitted 2024-04-16; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-05

CONDITIONS: Newly Diagnosed Type 1 Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: UCMSCs
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UCMSCs — Peripheral intravenous infusion of umbilical cord mesenchymal stem cells
  Arms: Experimental
Drug: Placebo — Peripheral intravenous infusion of Placebo
  Arms: Placebo Comparator

SUMMARY:
The aim is to investigate the safety and tolerability of intravenous infusion of allogeneic umbilical cord mesenchymal stem cells in pediatric patients diagnosed with newly onset type 1 diabetes

DETAILED DESCRIPTION:
This is an IIT study, where the first part is an open, dose escalating study consisting of 9 patients, 8-18 years of age. The second part is a randomized, double-blinded, placebo-controlled, IIT study in parallel design comparing allogeneic UCMSCs treatment to placebo in pediatric patients diagnosed with newly onset type 1 diabetes. Besides safety, preservation of endogenous insulin production (measured as C-peptide concentrations) together with metabolic control, diabetes treatment satisfaction and immunological profile will be assessed.

A total number of 24 patients will be enrolled in the study and followed for one year after UCMSCs/placebo treatment. Patients 8-18 years of age, both male and female, diagnosed for type 1 diabetes will be eligible. Providing informed consent and fulfillment of inclusion criteria and no exclusion criteria, they will within 6 months of diagnosis be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for diabetes according to the World Health Organization (WHO) guidelines from 1999.
2. Presence of at least one pancreatic autoantibody, or idiopathic type 1 diabetes mellitus (T1DM) with negative autoantibody testing.
3. Ages 8 to 18 years, regardless of gender.
4. Newly diagnosed T1DM within the past 6 months.
5. Fasting C-peptide ≥0.1 nmol/L and postprandial 2-hour C-peptide >0.2 nmol/L.
6. Voluntary acceptance of stem cell transplantation therapy by the individual, their family members, or legal guardians, and signing of an informed consent form.

Exclusion Criteria:

1. Diabetic ketoacidosis is not under control.
2. Severe allergic constitution.
3. BMI <14 or >35.
4. History of other autoimmune diseases, hematologic disorders.
5. HIV positive, carrier of viral hepatitis, active phase of viral hepatitis, or other uncontrolled infectious diseases.
6. History of acute pancreatitis, pulmonary embolism, or other thrombotic diseases, as well as severe diseases of the heart, liver, kidneys, respiratory system, nervous system, etc.
7. Suffering from gestational diabetes, monogenic diabetes, diabetes caused by pancreatic injury, or other secondary diabetes (such as Cushing's syndrome, thyroid dysfunction, or acromegaly-induced diabetes);
8. Pregnancy or planning pregnancy within 3 months before or after treatment, as well as breastfeeding women.
9. Mental illness, alcohol or drug abuse, inability to comply with treatment.
10. Known or suspected tumors.
11. According to the investigator's judgment, there are other clinical conditions that may endanger the safety of the subjects.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | Throughout the study until Week 52
  Changes in safety parameters of patients during the study period since baseline. Measured through the registration of adverse events and other safety parameters.
Efficacy Assessment | Week 52
  Delta-change of C-peptide Area Under the Curve (AUC) (0-120 min) for Mixed Meal Tolerance Test (MMTT) at Week 52 following UCMSCs/Placebo infusion when compared to test performed before start of treatment.

SECONDARY OUTCOMES:
Efficacy Assessment: HbA1c | Week 52
  Changes in patient HbA1c levels from baseline during the study period
Efficacy Assessment: Dose of exogenous insulin | Week 52
  Changes in daily exogenous insulin requirements during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yin, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided